CLINICAL TRIAL: NCT03865914
Title: Correlation Study Between Clinical Phenotype and Pathology of Type 2 Diabetic Nephropathy
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other); China-Japan Friendship Hospital (Other); Beijing Friendship Hospital (Other); Beijing Hospital (Other Government); Fourth Medical Center of PLA General Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Third Medical Center of PLA General Hospital (Unknown); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); Dongzhimen Hospital, Beijing (Other); Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xiangmei Chen, Professor,Chief physician,Academician of Chinese Academy of Engineering, Chinese PLA General Hospital
Other Study IDs: S2017-133-01
Record Dates: First submitted 2019-03-02; First posted 2019-03-07 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Diabetic Kidney Disease
Keywords: Diabetic kidney disease (DKD); Diabetic nephropathy（DN); non-diabetic renal diseases（ NDRD); Clinical-pathological correlations; differential diagnosis
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, kidney tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 diabetic nephropathy: The cohort will be followed for at least 10 years. The cohort will be divided into 2 groups according the pathological results of patients,and at least 3 groups according to clinical features such as renal function and proteinuria.

SUMMARY:
With the rapid increase of diabetic nephropathy worldwide, type 2 diabetes mellitus(DM) is the leading cause of end-stage renal disease(ESRD). Pathological types of diabetic kidney disease(DKD) could be mainly divided into diabetic nephropathy（DN）and non-diabetic renal diseases（NDRD）. There are no accurate renal biopsy indications and standardized operation procedures for type 2 diabetic nephropathy. The clinical stages of type 2 diabetic nephropathy still referred to the Mogensen stage of type 1 diabetic nephropathy. Thus, our study aim to clarify the differences in clinical phenotype between type 2 DN and type 2 NDRD, analysis the correlation between clinical and pathological features, and offer the criteria for clinical staging and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18, male or female
* Clinical diagnosed as type 2 diabetes mellitus
* The presence of renal impairment including: microalbuminuria or overt proteinuria or renal insufficiency
* The renal biopsy was performed with complete renal pathological diagnosis
* Obtaining the signed informed consent from patients

Exclusion Criteria:

* The history of the disease was not complete
* Clinical diagnosed as other secondary renal diseases
* Patients with hereditary kidney disease
* Autoimmune diseases
* Patients with malignant tumor were expected to survive less than 6 months
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The aim of this study is to clarify the differences in clinical phenotype between type 2 DN and type 2 NDRD, analysis the correlation between clinical and pathological features, and offer the criteria for clinical staging and prognosis.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-11-30 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
change in eGFR and urine protein from baseline | 24months
  eGFR is calculated using the CKD-EPI formula, involving gender, age, and serum creatinine.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangmei Chen, MD.&Ph.D, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The test has not been completed.

REFERENCES:
- [Derived] Dong Z, Wang X, Pan S, Weng T, Chen X, Jiang S, Li Y, Wang Z, Cao X, Wang Q, Chen P, Jiang L, Cai G, Zhang L, Wang Y, Yang J, He Y, Lin H, Wu J, Tang L, Zhou J, Li S, Li Z, Fu Y, Yu X, Geng Y, Zhang Y, Wang L, Xu M, Chen X. A multimodal transformer system for noninvasive diabetic nephropathy diagnosis via retinal imaging. NPJ Digit Med. 2025 Jan 24;8(1):50. doi: 10.1038/s41746-024-01393-1. PMID 39856403
- [Derived] Wang Q, Cheng H, Jiang S, Zhang L, Liu X, Chen P, Liu J, Li Y, Liu X, Wang L, Li Z, Cai G, Chen X, Dong Z. The relationship between diabetic retinopathy and diabetic nephropathy in type 2 diabetes. Front Endocrinol (Lausanne). 2024 Jan 26;15:1292412. doi: 10.3389/fendo.2024.1292412. eCollection 2024. PMID 38344659
- [Derived] Zhang W, Liu X, Dong Z, Wang Q, Pei Z, Chen Y, Zheng Y, Wang Y, Chen P, Feng Z, Sun X, Cai G, Chen X. New Diagnostic Model for the Differentiation of Diabetic Nephropathy From Non-Diabetic Nephropathy in Chinese Patients. Front Endocrinol (Lausanne). 2022 Jun 30;13:913021. doi: 10.3389/fendo.2022.913021. eCollection 2022. PMID 35846333
- [Derived] Qu YL, Dong ZY, Cheng HM, Liu Q, Wang Q, Yang HT, Mao YH, Li JJ, Liu HF, Geng YQ, Huang W, Liu WH, Xie HD, Peng F, Li S, Jiang SS, Li WZ, Duan SW, Feng Z, Zhang WG, Liu YN, Tian JZ, Chen XM. Evaluation of Renal Impairment in Patients with Diabetic Kidney Disease by Integrated Chinese and Western Medicine. Chin J Integr Med. 2023 Apr;29(4):308-315. doi: 10.1007/s11655-022-3520-0. Epub 2022 Jun 9. PMID 35679002